CLINICAL TRIAL: NCT03876366
Title: Fertility Preservation in Men Affected by Cancer: Assessment of Patients' Needs and Development of an Online Decision-aid
Brief Title: Fertility Preservation in Men Affected by Cancer
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-02069; sp19Tschudin
Record Dates: First submitted 2019-02-26; First posted 2019-03-15 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: cancer patients; male cancer patients; Decision Aid (DA); online Decision Aid tool
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: online survey — Part 1: online survey (quantitative) with questions on basic socio-demographic data, medical data and family characteristics (e.g. age, ethnicity, education) and information about FP.
Other: focus group meeting — Part 2: At the end of the online survey, participants are invited to attend one of the consecutively performed focus groups conducted according to standardized focus group methodology and moderated by a clinical psychologist and a specialist in reproductive medicine.

SUMMARY:
This is a single center cross-sectional retrospective study with a quantitative and qualitative approach (phase 1 and 2). In phase 1 an online survey will be realized and targets male cancer survivors. Phase 2 will take a qualitative approach, in which information about patient's experiences, needs and helpful support will be collected by establishing focus groups of cancer patients who had been diagnosed during the reproductive age.

In the end, the results of this study will be integrated into the development of an online support tool concerning Fertility Preservation (FP).

ELIGIBILITY:
Inclusion Criteria:

* German speaking
* Cancer diagnosis within the last 10 years (minimum age at diagnosis 13 years)
* Cancer therapy that was expected to impair fertility

Exclusion Criteria:

* Prepubertal at diagnosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who are/were possible candidates for FP (patients with fertility compromising cancer treatment) will be invited to participate. Eligible patients will be approached by their former or current treating oncologist, urologist or specialist in reproductive medicine.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
male cancer patients level of information with regard to FP | Phase 1 online survey at baseline
  Phase 1: exploratory online survey inquiring male cancer patients level of information with regard to FP
male cancer patients level of information with regard to FP | Phase 2 focus group meeting (approx. 2 to 4 weeks after baseline)
  Phase 2: interview (strictly exploratory) in focus groups collecting data on male cancer patients level of information with regard to FP

SECONDARY OUTCOMES:
male cancer patients needs regarding decision-making about FP | Phase 1 online survey at baseline
  exploratory online survey inquiring which kind of support regarding decision-making about FP do male cancer patients consider helpful
male cancer patients expectation with regard to an online DA tool about FP | Phase 1 online survey at baseline
  exploratory online survey inquiring how an online Decision Aid (DA) tool about FP has to be designed in order to be helpful for male cancer patients
male cancer patients needs regarding decision-making about FP | Phase 2 focus group meeting (approx. 2 to 4 weeks after baseline)
  Phase 2: interview (strictly exploratory) in focus groups evaluating which kind of support regarding decision-making about FP male cancer patients consider helpful
male cancer patients expectation with regard to an online DA tool about FP | Phase 2 focus group meeting (approx. 2 to 4 weeks after baseline)
  Phase 2: interview (strictly exploratory) in focus groups evaluating how an online DA tool about FP has to be designed in order to be helpful for male cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Sibil Tschudin, PD Dr. med, Principal Investigator — Frauenklinik Universitätsspital Basel
Locations (1):
- Frauenklinik University Hospital Basel, Basel, Switzerland